CLINICAL TRIAL: NCT06231433
Title: Effect of Factional CO2 Laser Treatment on Vaginal Symptoms and Sexual Dysfunction in Women With Systemic Sclerosis
Brief Title: Effects of Fractional CO2 Laser Treatment on Vaginal Symptoms and Sexual Dysfunction in Women With Systemic Sclerosis
Acronym: SCLERDERMCO2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Salvatore, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCLERODERMCO2
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Systemic Sclerosis; Vulvovaginal Signs and Symptoms; Sexual Function Disturbances
MeSH Terms: conditions — Scleroderma, Systemic; Sexual Dysfunctions, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women affected by Systemic Sclerosis and vulvovaginal atrophy (Experimental): CO2 vaginal laser
  Interventions: Device: CO2 Vaginal Laser

INTERVENTIONS:
Device: CO2 Vaginal Laser — CO2 Vaginal laser

SUMMARY:
Women affected by Systemic Sclerosis and Vulvovaginal Atrophy will be submitted to a cycle composed of five vaginal CO2 laser treatment (SmartXide2 V2LR, Monalisa Touch, DEKA, Florence, Italy - Hi Scan V2LR con sonda vaginale a 360 °, dot power 30 watt, dwell time 1000 μs, dot spacing 1000 μm smart stack 1-3, emission mode deka pulse) every 30-40 days.

At 1-month follow up from the last vaginal laser treatment (6 months from baseline) vagina and sexual health will be assessed by a 1-5 Likert scale, a 0-10 Visual Analogue Scale for vulvovaginal symptoms and the Female Sexual Function Index.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Systemic Sclerosis; - vulvovaginal symptoms

Exclusion Criteria:

* gynecological neoplasia; - pregnancy; - pelvic organ prolapse; - vaginal and urinary infection; - pudendal neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
1-5 Likert Scale | Six months follow up
  Scale of satisfaction for the treatment

SECONDARY OUTCOMES:
0-10 Visual Analogue Scale | Six months follow up
  Scale of vulvovaginal symptoms severity
Female Sexual Function Index | Six months follow up
  Questionnaire assessing sexual function

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No